CLINICAL TRIAL: NCT03565744
Title: The B'N Fit POWER Initiative: A School-Based Wellness Initiative for Bronx Youth
Acronym: BNFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-5917
Record Dates: First submitted 2018-05-02; First posted 2018-06-21 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Overweight and Obesity
Keywords: obesity; adolescents; school-based; weight management; wellness
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a quasi-experimental trial of B'N Fit POWER in two middle schools that have both an onsite MSHP and MMCC service.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - B'N Fit POWER (Experimental): Participants enrolling in B'N Fit POWER afterschool program will be assigned to Group 1.
  Interventions: Behavioral: B'N Fit POWER
- Group 2 - Standard of Care (No Intervention): All other PS/MS-95 participants who completed the screening (approximately 50) will be in comparison Group 2
- Group 3 - Standard of Care (No Intervention): Participants at an additional school site completing the screening (approximately 100) will be in an additional comparison Group 3.

INTERVENTIONS:
Behavioral: B'N Fit POWER — Participants will undergo a medical assessment and using an Electronic Medical Record (EMR) template, providers will screen for a healthy weight and the 7 target behaviors. Participants will set goals with the provider to attain one of the target behaviors and will receive an EMR-generated treatment plan summarizing healthy weight and target behavior goals. At 20-minute follow-up visits during the school day, the provider will review weight and target behavior attainment and monitor co-morbidities and barriers to participation. Group 1 participants will also have access to daily MMCC afterschool programming from 3-6pm from September through May each year with tailored programming including weekly core nutrition, behavior, and cooking classes and at least five hours of physical activity.
  Arms: Group 1 - B'N Fit POWER

SUMMARY:
The findings of this study will establish the feasibility and efficacy of B'N Fit POWER and given the wide presence of MSHP, MMCC and other afterschool programs, there is significant potential for dissemination of B'N Fit POWER to many other clinic-community partnership sites enabling the development of a larger grant that will test the effectiveness and dissemination process to several schools in the Bronx. The translation of a traditional clinical-based weight-loss intervention to adapting and implementing such an intervention in a real-world school setting is more relevant and sustainable for advancing a culture of health and promoting diabetes risk reduction in Bronx youth.

DETAILED DESCRIPTION:
In this proposal, the investigators aim to test a school-based intervention to promote resilience and prevent obesity related co-morbidities for impoverished racial/ethnic minority Bronx youth who are at increased risk for diabetes. B'N Fit POWER is a wellness program that integrates existing school wellness promotion activities, the Montefiore School Health Program (MSHP) - a network of school-based health clinics, and the Mosholu Montefiore Community Center (MMCC) - a network of afterschool programming, to promote health and build on the resilience of the adolescents. It offers culturally-relevant guidance related to the attainment of 7 Target Behaviors, namely to increase fruit, vegetable and sugar-free beverage intake, obtain adequate sleep, daily physical activity, eating breakfast and lunch daily, and limiting fast food and unhealthy snacks. Although B'N Fit POWER targets youth with overweight and obesity and at high risk for diabetes, it is open to all middle school students at the school, via community-led recruitment efforts to reduce obesity-related stigma by promoting wellness and fitness. Grounded in Youth Development (YD) Theory and using the principles of Community Based Participatory Research (CBPR) the program integrates patient, family, clinical, and community linkages, and targets individual behaviors as well as the school environment to address environmental and structural barriers to behavioral change. YD program elements are incorporated to build positive identity, youth resilience, and foster youth leadership by having youth contribute to planning community activities with incentives to promote attendance and retention. The investigators will conduct a quasi-experimental trial of B'N Fit POWER and will compare participants receiving B'N Fit POWER (Group 1) to two comparison groups: one from the same school receiving standard of care (Group 2) and, to assess the external validity of Group 2 in terms of characteristics and outcomes, an additional group from another school also receiving standard of care (Group 3) to address the following specific aims: 1) Determine whether B' N Fit POWER is effective in improving fitness, healthy weight attainment, and 7 target behaviors; 2) To assess the impact of moving the B'N Fit program into a school setting on participant engagement; and 3) To assess the mediating pathways associated with program effects. Following an initial health screening, participants enrolling in B'N Fit POWER (Group 1) will receive comprehensive medical assessments at the MSHP integrated with MMCC afterschool programming that incorporates a curriculum focusing on 7 Target Behaviors during weekly leadership sessions and daily physical activity. The comparison groups receive the standard of care (standard MSHP and MMCC afterschool program). Effects of the program will be evaluated using data routinely collected at the schools (e.g. anthropometrics and labs from clinic and the school fitnessgram, attendance, grades) and surveys. Multivariate logistic regressions and mixed-effects linear models will assess program effects for categorical or continuous outcomes and the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) approach will identify barriers and solutions to implementation.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 and no older than 14 when recruited at baseline
* A parent or guardian will be available in person or by phone at all clinical visits.
* Registered in both the Montefiore School Health Program clinic and Mosholu Montefiore Community Health Center afterschool program at Public School (PS) /Middle School (MS) 95

Exclusion Criteria:

* Has a major mental illness that would render them incapable of consenting for the research or complying with the B'N Fit POWER afterschool program protocol
* Has medical problems that make it unsafe for them to participate in the afterschool program.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change in BMI | baseline, 4 -7 months, 8 - 10 months, 11 - 12 months, 12 - 13 months (final visit)
  height (in m) and weight (in kg) will be combined to report BMI in kg/m^2. Visit schedule: Time 1) Baseline June screen; Time 2) 1st clinic visit from Sept. - Dec.; Time 3) 2nd clinic visit from Jan.-March; Time 4) 3rd clinic visit from April-May; Time 5) Final June screen

SECONDARY OUTCOMES:
Change in cardiovascular disease risk | 4 -7 months (baseline clinic visit), 11 - 12 months (final clinic visit) if abnormal during the baseline clinic visit
  (LDL-cholesterol, triglycerides, and HDL-cholesterol will be measured). Visit schedule: Time 2) 1st clinic visit from Sept. - Dec.; Time 4) third and final clinic visit from April-May
Change in diabetes risk | 4 -7 months (baseline clinic visit), 11 - 12 months (final clinic visit) if abnormal during the baseline clinic visit
  HgBA1C will be measured as a marker of insulin resistance. Visit schedule: Time 2) 1st clinic visit from Sept. - Dec.; Time 4) third and final clinic visit from April-May
Change in nutrition and physical activity knowledge | baseline, 12 - 13 months (final visit)
  B'N Fit Survey includes questions assessing nutrition and physical activity knowledge. Visit schedule: Time 1) Baseline June screen; Time 5) Final June screen
Change in school attendance and performance | baseline, 12 - 13 months (final visit)
  B'N Fit Survey includes questions assessing school attendance and performance.Visit schedule: Time 1) Baseline June screen; Time 5) Final June screen
Change in target behaviors | Time Frame: baseline, 4 -7 months, 8 - 10 months, 11 - 12 months, 12 - 13 months (final visit)
  Target behavior survey assesses number of daily fruit, vegetable, sugar-free beverage, and sugary beverage servings consumed, daily hours of sleep, number of hours of physical activity on a weekly basis, number of days that breakfast and lunch are eaten daily, number of days that fast food and unhealthy snacks are consumed. Visit schedule: Time 1) Baseline June screen; Time 2) 1st clinic visit from Sept. - Dec.; Time 3) 2nd clinic visit from Jan.-March; Time 4) 3rd clinic visit from April-May; Time 5) Final June screen
Change in fitness | baseline, 12 - 13 months (final visit)
  Fitness will be assessed by measuring cardiovascular fitness, abdominal strength, trunk strength, arm strength and flexibility by the routinely collected NYC FITNESSGRAM. Visit schedule: Time 1) Baseline June screen; Time 5) Final June screen
Program attendance | Clinic attendance: 4 -7 months, 8 - 10 months, 11 - 12 months; Afterschool attendance: 4-13 months
  Attendance at clinic sessions and afterschool program sessions. Visit Schedule: 1) 1st fall clinic visit (Time 2); 2) 2nd winter clinic visit (Time 3); 3) 3rd spring clinic visit (Time 4) ; 4) Daily attendance for 10 months that afterschool is in session

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Walker, PhD, RN, Study Director — Albert Einstein College of Medicine; Jessica Rieder, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- PS-95, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Yamron E, Moon JY, Meissner P, Wylie-Rosett J, Shankar V, Rieder J. Trends in health behavior at an afterschool program: the impact of COVID-19 on students' behavior. Res Sq [Preprint]. 2023 Mar 28:rs.3.rs-2679660. doi: 10.21203/rs.3.rs-2679660/v1. PMID 37034787
- [Result] Rieder J, Cain A, Carson E, Benya A, Meissner P, Isasi CR, Wylie-Rosett J, Hoffman N, Kelly C, Silver EJ, Bauman LJ. Pilot Project to Integrate Community and Clinical Level Systems to Address Health Disparities in the Prevention and Treatment of Obesity among Ethnic Minority Inner-City Middle School Students: Lessons Learned. J Obes. 2018 Mar 26;2018:6983936. doi: 10.1155/2018/6983936. eCollection 2018. PMID 29850232
- [Result] Rieder J, Moon JY, Joels J, Shankar V, Meissner P, Johnson-Knox E, Frohlich B, Davies S, Wylie-Rosett J. Trends in health behavior and weight outcomes following enhanced afterschool programming participation. BMC Public Health. 2021 Apr 7;21(1):672. doi: 10.1186/s12889-021-10700-4. PMID 33827501